CLINICAL TRIAL: NCT02798913
Title: Effects of Prolonged Dual Antiplatelet Therapy With Clopidogrel Plus Acetylsalicylic Acid (ASA) After Percutaneous Lower Extremity Revascularization in Patients With Peripheral Arterial Disease
Brief Title: Effects of Prolonged DAPT After Lower Extremity Percutaneous Transluminal Angioplasty (PTA) in Patients With LE-PAD
Acronym: LONGDAPTPAD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Giuseppe Giugliano, MD, PhD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 103/13
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Peripheral Artery Disease
Keywords: dual antiplatelet therapy; peripheral transluminal angioplasty
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short DAPT (Experimental): Patients who will be treated after PTA with acetylsalicylic acid 100 mg/day life-long + clopidogrel 75 mg/day for 3 months
  Interventions: Drug: Short DAPT
- Long DAPT (Experimental): Patients who will be treated after PTA with acetylsalicylic acid 100 mg/day life-long + clopidogrel 75 mg/day for 12 months
  Interventions: Drug: Long DAPT

INTERVENTIONS:
Drug: Short DAPT — acetylsalicylic acid 100 mg/day life-long + clopidogrel 75 mg/day for 3 months
  Other Names: 3 months ASA + Clopidogrel
  Arms: Short DAPT
Drug: Long DAPT — acetylsalicylic acid 100 mg/day life-long + clopidogrel 75 mg/day for 12 months
  Other Names: 12 months ASA + Clopidogrel
  Arms: Long DAPT

SUMMARY:
The objective of the present study was to evaluate the prognostic impact of prolonged dual antiplatelet therapy (DAPT) with acetylsalicylic acid plus clopidogrel on the incidence of major adverse cardiovascular events and major adverse limb events after percutaneous lower extremity revascularization in patients with lower extremity peripheral arterial disease (LE-PAD).

ELIGIBILITY:
Inclusion Criteria:

* LE-PAD at stage 2 of Fontaine's classification (intermittent claudication)
* successful PTA of aorto-iliac, femoro-popliteal ore below-the-knee segments

Exclusion Criteria:

* critical limb ischemia
* recent acute coronary syndrome (< 12 months)
* recent cerebrovascular event (< 12 months)
* recent myocardial, carotid or peripheral revascularization (< 12 months)
* recent history of bleeding (< 12 months)
* other indication for clopidogrel therapy
* indication for anticoagulation
* de-compensated heart failure
* malignant neoplasm

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Events + incidence of Major Adverse Limb Events | 24 months post-PTA
  Impact of prolonged vs. short dual antiplatelet therapy after PTA on the incidence of major adverse cardiovascular events (death from cardiovascular cause, myocardial infarction, stroke, coronary or carotid revascularization) + the incidence of major adverse limb events (restenosis, occlusion, or new revascularization of target lesion, new stenosis, occlusion, or revascularization of not-target lesion, onset of acute and critical limb ischemia, amputation).

SECONDARY OUTCOMES:
Incidence of minor and major bleedings according to the GUSTO classification | 24 months post-PTA
  Incidence of minor and major bleedings according to the Global Utilization of Streptokinase and Tissue plasminogen activator for Occluded coronary arteries classification

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Trimarco, Study Director — Federico II University; Giovanni Esposito, MD, PhD, Principal Investigator — Federico II University
Locations (1):
- Department of Advanced Biomedical Sciences, University of Naples "Federico II", Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Antithrombotic Trialists' Collaboration. Collaborative meta-analysis of randomised trials of antiplatelet therapy for prevention of death, myocardial infarction, and stroke in high risk patients. BMJ. 2002 Jan 12;324(7329):71-86. doi: 10.1136/bmj.324.7329.71. PMID 11786451
- [Background] CAPRIE Steering Committee. A randomised, blinded, trial of clopidogrel versus aspirin in patients at risk of ischaemic events (CAPRIE). CAPRIE Steering Committee. Lancet. 1996 Nov 16;348(9038):1329-39. doi: 10.1016/s0140-6736(96)09457-3. PMID 8918275
- [Background] Belch JJ, Topol EJ, Agnelli G, Bertrand M, Califf RM, Clement DL, Creager MA, Easton JD, Gavin JR 3rd, Greenland P, Hankey G, Hanrath P, Hirsch AT, Meyer J, Smith SC, Sullivan F, Weber MA; Prevention of Atherothrombotic Disease Network. Critical issues in peripheral arterial disease detection and management: a call to action. Arch Intern Med. 2003 Apr 28;163(8):884-92. doi: 10.1001/archinte.163.8.884. No abstract available. PMID 12719196
- [Background] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group; Bell K, Caporusso J, Durand-Zaleski I, Komori K, Lammer J, Liapis C, Novo S, Razavi M, Robbs J, Schaper N, Shigematsu H, Sapoval M, White C, White J, Clement D, Creager M, Jaff M, Mohler E 3rd, Rutherford RB, Sheehan P, Sillesen H, Rosenfield K. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). Eur J Vasc Endovasc Surg. 2007;33 Suppl 1:S1-75. doi: 10.1016/j.ejvs.2006.09.024. Epub 2006 Nov 29. No abstract available. PMID 17140820
- [Background] European Stroke Organisation; Tendera M, Aboyans V, Bartelink ML, Baumgartner I, Clement D, Collet JP, Cremonesi A, De Carlo M, Erbel R, Fowkes FG, Heras M, Kownator S, Minar E, Ostergren J, Poldermans D, Riambau V, Roffi M, Rother J, Sievert H, van Sambeek M, Zeller T; ESC Committee for Practice Guidelines. ESC Guidelines on the diagnosis and treatment of peripheral artery diseases: Document covering atherosclerotic disease of extracranial carotid and vertebral, mesenteric, renal, upper and lower extremity arteries: the Task Force on the Diagnosis and Treatment of Peripheral Artery Diseases of the European Society of Cardiology (ESC). Eur Heart J. 2011 Nov;32(22):2851-906. doi: 10.1093/eurheartj/ehr211. Epub 2011 Aug 26. No abstract available. PMID 21873417
- [Background] Yusuf S, Zhao F, Mehta SR, Chrolavicius S, Tognoni G, Fox KK; Clopidogrel in Unstable Angina to Prevent Recurrent Events Trial Investigators. Effects of clopidogrel in addition to aspirin in patients with acute coronary syndromes without ST-segment elevation. N Engl J Med. 2001 Aug 16;345(7):494-502. doi: 10.1056/NEJMoa010746. PMID 11519503
- [Background] Chen ZM, Jiang LX, Chen YP, Xie JX, Pan HC, Peto R, Collins R, Liu LS; COMMIT (ClOpidogrel and Metoprolol in Myocardial Infarction Trial) collaborative group. Addition of clopidogrel to aspirin in 45,852 patients with acute myocardial infarction: randomised placebo-controlled trial. Lancet. 2005 Nov 5;366(9497):1607-21. doi: 10.1016/S0140-6736(05)67660-X. PMID 16271642
- [Background] Mauri L, Kereiakes DJ, Normand SL, Wiviott SD, Cohen DJ, Holmes DR, Bangalore S, Cutlip DE, Pencina M, Massaro JM. Rationale and design of the dual antiplatelet therapy study, a prospective, multicenter, randomized, double-blind trial to assess the effectiveness and safety of 12 versus 30 months of dual antiplatelet therapy in subjects undergoing percutaneous coronary intervention with either drug-eluting stent or bare metal stent placement for the treatment of coronary artery lesions. Am Heart J. 2010 Dec;160(6):1035-41, 1041.e1. doi: 10.1016/j.ahj.2010.07.038. PMID 21146655
- [Background] Mehta SR, Yusuf S, Peters RJ, Bertrand ME, Lewis BS, Natarajan MK, Malmberg K, Rupprecht H, Zhao F, Chrolavicius S, Copland I, Fox KA; Clopidogrel in Unstable angina to prevent Recurrent Events trial (CURE) Investigators. Effects of pretreatment with clopidogrel and aspirin followed by long-term therapy in patients undergoing percutaneous coronary intervention: the PCI-CURE study. Lancet. 2001 Aug 18;358(9281):527-33. doi: 10.1016/s0140-6736(01)05701-4. PMID 11520521
- [Background] James SK, Roe MT, Cannon CP, Cornel JH, Horrow J, Husted S, Katus H, Morais J, Steg PG, Storey RF, Stevens S, Wallentin L, Harrington RA; PLATO Study Group. Ticagrelor versus clopidogrel in patients with acute coronary syndromes intended for non-invasive management: substudy from prospective randomised PLATelet inhibition and patient Outcomes (PLATO) trial. BMJ. 2011 Jun 17;342:d3527. doi: 10.1136/bmj.d3527. PMID 21685437
- [Background] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Background] Grines CL, Bonow RO, Casey DE Jr, Gardner TJ, Lockhart PB, Moliterno DJ, O'Gara P, Whitlow P; American Heart Association; American College of Cardiology; Society for Cardiovascular Angiography and Interventions; American College of Surgeons; American Dental Association; American College of Physicians. Prevention of premature discontinuation of dual antiplatelet therapy in patients with coronary artery stents: a science advisory from the American Heart Association, American College of Cardiology, Society for Cardiovascular Angiography and Interventions, American College of Surgeons, and American Dental Association, with representation from the American College of Physicians. Circulation. 2007 Feb 13;115(6):813-8. doi: 10.1161/CIRCULATIONAHA.106.180944. Epub 2007 Jan 15. PMID 17224480
- [Background] Visona A, Tonello D, Zalunardo B, Irsara S, Liessi G, Marigo L, Zotta L. Antithrombotic treatment before and after peripheral artery percutaneous angioplasty. Blood Transfus. 2009 Jan;7(1):18-23. doi: 10.2450/2008.0008-08b. No abstract available. PMID 19290075
- [Background] Tepe G, Bantleon R, Brechtel K, Schmehl J, Zeller T, Claussen CD, Strobl FF. Management of peripheral arterial interventions with mono or dual antiplatelet therapy--the MIRROR study: a randomised and double-blinded clinical trial. Eur Radiol. 2012 Sep;22(9):1998-2006. doi: 10.1007/s00330-012-2441-2. Epub 2012 May 10. PMID 22569995
- [Background] Dorffler-Melly J, Koopman MM, Prins MH, Buller HR. Antiplatelet and anticoagulant drugs for prevention of restenosis/reocclusion following peripheral endovascular treatment. Cochrane Database Syst Rev. 2005 Jan 25;(1):CD002071. doi: 10.1002/14651858.CD002071.pub2. PMID 15674891
- [Background] Belch JJ, Dormandy J; CASPAR Writing Committee; Biasi GM, Cairols M, Diehm C, Eikelboom B, Golledge J, Jawien A, Lepantalo M, Norgren L, Hiatt WR, Becquemin JP, Bergqvist D, Clement D, Baumgartner I, Minar E, Stonebridge P, Vermassen F, Matyas L, Leizorovicz A. Results of the randomized, placebo-controlled clopidogrel and acetylsalicylic acid in bypass surgery for peripheral arterial disease (CASPAR) trial. J Vasc Surg. 2010 Oct;52(4):825-33, 833.e1-2. doi: 10.1016/j.jvs.2010.04.027. Epub 2010 Aug 1. PMID 20678878
- [Background] GUSTO investigators. An international randomized trial comparing four thrombolytic strategies for acute myocardial infarction. N Engl J Med. 1993 Sep 2;329(10):673-82. doi: 10.1056/NEJM199309023291001. PMID 8204123